CLINICAL TRIAL: NCT02616913
Title: A Single Dose, Double Blind, Randomized, Crossover Placebo- and Moxifloxacin (Open Label)-Controlled Study to Evaluate the Cardiac Effects of a Novel Food Ingredient in Healthy Male Subjects
Brief Title: Evaluation of the Cardiac Effects of a Novel Food Ingredient in Healthy Male Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Collaborators: Ajinomoto Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 8280290
Record Dates: First submitted 2015-11-05; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Cardiovascular Abnormalities
MeSH Terms: conditions — Cardiovascular Abnormalities | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- R,R-monatin (Experimental): 150 mg single dose
  Interventions: Other: R,R-monatin
- Moxifloxacin (Active Comparator): 400 mg tablet single dose
  Interventions: Other: Moxifloxacin
- Placebo (Placebo Comparator): placebo single dose
  Interventions: Other: Placebo

INTERVENTIONS:
Other: R,R-monatin — Each subject consumes test article R,R-monatin (150 mg) in one of 3 treatment periods
  Arms: R,R-monatin
Other: Moxifloxacin — Each subject consumes moxifloxacin (400 mg; positive control) in one of 3 treatment periods
  Arms: Moxifloxacin
Other: Placebo — Each subject consumes placebo in one of 3 treatment periods
  Arms: Placebo

SUMMARY:
This study evaluates if a single oral dose of 150 mg of the novel food ingredient (AME001, R,R-monatin) does not have an effect on the Fridericia-corrected QT ECG interval (QTcF) exceeding 10 milliseconds (msec). Each subject will consume test article (150 mg), placebo, and moxifloxacin (400 mg; positive control) in each of 3 treatment periods.

DETAILED DESCRIPTION:
This study is specifically designed to evaluate the potential effects of ingestion of the novel food ingredient on cardiac safety. The objective will be fulfilled by assessing cardiac parameters including heart rate, blood pressure, and ECG/QT interval in healthy adult male subjects following a single dose oral administration of the test article.

The primary objective of this study is to demonstrate that a single oral dose of 150 mg of the test article does not have an effect on the Fridericia-corrected QT ECG interval (QTcF) exceeding 10 milliseconds (msec).

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking healthy male between 18 and 45 years of age;
* BMI within the range 18.0 to 30.0 kg/m2, inclusive, and with a body weight ≥60 kg;
* Subjects with a partner of childbearing potential agree to use dual methods of contraception from Check-in until 3 months (90 days) after the last treatment, and to provide no sperm donation from Check-in until 3 months (90 days) after last administration of test article. Double barrier methods include: a male condom with spermicide; a sterile sexual partner; use by female sexual partner of an intrauterine device (IUD) with spermicide; a female condom with spermicide; contraceptive sponge with spermicide; an intravaginal system (e.g. NuvaRing®) a diaphragm with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives;
* Subjects must be in good health, determined by no clinically significant or relative abnormalities identified by medical history, full physical examination, vital signs measurements, 12-lead ECG, and clinical laboratory evaluations;
* Subjects must be willing and able to comply with all study requirements;
* Subjects must have given written informed consent.

Exclusion Criteria:

* Presence of history of any disorder that may prevent successful completion of the study, in the opinion of the investigator;
* Subjects who have received an investigational product (investigational pharmaceutical or a medical device) within the 30 days prior to Day -1 of the first treatment period (Check-in);
* Any cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease that are clinically significant in the opinion of the Investigator;
* Any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of test article (cholecystectomy and appendectomy allowed);
* Any acute disease state (e.g. nausea, vomiting, fever, or diarrhea) within 7 days before Day -1 of the first treatment period (Check-in);
* History of drug abuse within 1 year before Day -1 of the first treatment period, as assessed by the Investigator, where drug abuse is defined as: recurrent use of a substance resulting in failure to fulfill a person's major role obligation at work or at home; recurrent use in physically hazardous situations; recurrent substance-related legal problems; or continued use despite persistent or recurrent social or interpersonal problems caused or exacerbated by the substance;
* Admitted alcohol abuse or history of alcohol use that may interfere with the subject's ability to comply with the protocol requirements in the opinion of the Investigator;
* Family history of Long QT Syndrome and/or unexplained sudden cardiac death;
* Any clinically important deviation from normal limits in physical examination, vital signs, 12-lead ECG, or clinical laboratory test results, in the opinion of the Investigator;
* Electrolyte results for Ca, Mg, and K outside of normal limits; all other electrolytes will be assessed by the Investigator for clinical significance and subjects will be excluded if results are deemed clinically significant;
* QTc duration ≥450 msec based on machine-read tracing at Screening. Recalculation into QTcF and up to 1 repeat may be allowed; further repeats may be allowed if discussed and agreed with the Medical Monitor;
* Positive serologic findings for HIV antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies;
* Positive findings on urine drug screen (e.g. amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates);
* History of any clinically important allergy to moxifloxacin;
* History of any significant adverse drug reaction to any fluoroquinolone;
* Use of any investigational medications within 30 days prior to the first dose and the use of any prescription medications during the interval from 14 days prior to Check-in for the first treatment period until after the completion of the study. In addition, subjects will refrain from the use of any over-the-counter non-prescription medications (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations; except for the occasional use of acetaminophen), and all dietary supplements, within 7 days before Day -1 of the first treatment period (Check-in);
* Consumption of any caffeine-containing products (e.g. coffee, tea, chocolate, or soda) or alcoholic beverages within 72 hours before Day -1 of the first treatment period (Check-in).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Fridericia-corrected QT ECG interval (QTcF) | 24 hours

SECONDARY OUTCOMES:
Electrocardiogram parameters: Heart rate, PR interval, QRS and T-wave morphology | 24 hours